CLINICAL TRIAL: NCT04260633
Title: Optimizing Aligner Wear Time and Change Frequency: A Single-Blind, Randomized Control Trial
Brief Title: Optimizing Aligner Wear Time and Change Frequency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harvard School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB19-0644
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Adjunctive Usage of Vibrational Therapy; Dental Monitoring Accuracy

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, randomized, controlled, single-blind, parallel group clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (No Intervention): 22-hour tray wear time, DM assisted aligner change frequency
- Group 2 (Active Comparator): 22-hour tray wear time, VPro+ (active), DM assisted aligner change frequency
  Interventions: Device: Dental Monitoring assisted aligner change, 12-hour tray wear time and VPro+ are the interventions for the trial.
- Group 3 (Sham Comparator): 22-hour tray wear time, VPro+ (inactive), DM assisted aligner change frequency
  Interventions: Device: Dental Monitoring assisted aligner change, 12-hour tray wear time and VPro+ are the interventions for the trial.
- Group 4 (Active Comparator): 12-hour tray wear time, VPro+ (active), DM assisted aligner change frequency
  Interventions: Device: Dental Monitoring assisted aligner change, 12-hour tray wear time and VPro+ are the interventions for the trial.
- Group 5 (Sham Comparator): 12-hour tray wear time, VPro+ (inactive), DM assisted aligner change frequency
  Interventions: Device: Dental Monitoring assisted aligner change, 12-hour tray wear time and VPro+ are the interventions for the trial.

INTERVENTIONS:
Device: Dental Monitoring assisted aligner change, 12-hour tray wear time and VPro+ are the interventions for the trial. — The current standard of care for clear aligner use as suggested by Invisalign is unclear as to how frequently aligners should be changed. We suspect that the frequency for aligner change as determined by the orthodontist using Dental Monitoring will be variable for every participant.
  Vpro+ is an adjunctive therapeutic tool for clear aligner treatment. It is proposed to deliver high frequency vibrations to reduce treatment time and pain associated with clear aligners.
  Align Technology suggests 22-hour wear time for clear aligner therapy. Participants in two arms of the study will be asked to wear the trays for about half the recommended wear time to assess whether night-time aligner wear will be sufficient for successful treatment.
  Arms: Group 2; Group 3; Group 4; Group 5

SUMMARY:
This study aims to help improve individualization and optimization of clear aligner therapy through the use of new technologies in orthodontics. The study will compare 12-hour and 22-hour tray wear time and evaluate the adjunctive use of Vpro+. The study clinicians will use Dental Monitoring to monitor study participants throughout the trial and will use the Dental Monitoring system to instruct patients to continue or stay on their clear aligners. The outcome of the study will be the time it takes to complete 10 trays.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18-65 years of age with complete adult dentition, with Class I malocclusion or mild Class II/III malocclusions who are currently in treatment.
* Subjects who do not have systemic diseases that affect orthodontic tooth movement such as patients who are using hormone replacement medications, bone diseases such as osteoporosis or hyper/hypo-thyroidism
* Periodontal probing depths (PD) < 4mm, gingival index (GI) ≤1, and plaque index (PI) ≤1
* Patients currently in orthodontic treatment with Invisalign who are currently changing their trays every 7 - 10 days
* Participant must have a smartphone that is capable of downloading and storing the Dental Monitoring application
* Participants must be able to master the use of the Dental Monitoring Application

Exclusion Criteria:

Inclusion:

* Male and female subjects ages 18-65 years of age with complete adult dentition, with Class I malocclusion or mild Class II/III malocclusions who are currently in treatment.
* Subjects who do not have systemic diseases that affect orthodontic tooth movement such as patients who are using hormone replacement medications, bone diseases such as osteoporosis or hyper/hypo-thyroidism
* Periodontal probing depths (PD) < 4mm, gingival index (GI) ≤1, and plaque index (PI) ≤1
* Patients currently in orthodontic treatment with Invisalign who are currently changing their trays every 7 - 10 days
* Participant must have a smartphone that is capable of downloading and storing the Dental Monitoring application
* Participants must be able to master the use of the Dental Monitoring Application

Exclusion:

* Subjects who have within the last 6 mo taken any antibiotic medications or have had any periodontal treatments
* Subjects who have taken/are taking medications that affect bone remodeling: anti-resorptive medications, medications that may affect hormone levels, thyroid replacement medications, corticosteroids, and daily nonsteroidal anti-inflammatory medications
* Subjects who have had chemotherapy or radiation therapy in the last 6 mo
* Subjects who present with severe class II/III malocclusions
* Subjects who present with class I malocclusions but have severe crowding (> 7 mm) that requires extraction, >4 mm positive overjet and > 2 mm negative overjet, extreme deep bite ( > 90%), severe open bite (>2 mm)
* Women who are pregnant
* Patients that smoke
* Patients with active caries
* Patients that require interproximal reduction or attachments in the remaining prescription
* Patients who have temporary anchorage devices in place
* Patients who have vertigo or issues with their temporomandibular joint
* Patients with less than 3 mo. remaining in aligner treatment
* Patients who have documented bruxism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to complete 10 trays to determine the average aligner change frequency measured at the completion of the study | 70-140 days